CLINICAL TRIAL: NCT04298437
Title: Optimizing Treatment for Parents of Children With Emotional and Behavioural Problems (OPTED)
Brief Title: Addressing Depression and Positive Parenting Techniques (ADAPT)
Acronym: ADAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 028/2019
Record Dates: First submitted 2020-02-21; First posted 2020-03-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Depression; Emotional Problem; Disruptive Behavior Disorder; Attention Deficit Hyperactivity Disorder; Conduct Disorder; Oppositional Defiant Disorder; Behavior Problem
Keywords: Depression; Emotional and Behavioural Difficulties; Disruptive Behaviour Disorders; Oppositional Defiant Disorder; Dialectical Behaviour Therapy; Parenting Skills; Behavioural Parenting Training; Conduct Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Depression; Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder with Hyperactivity; Conduct Disorder; Oppositional Defiant Disorder; Mental Disorders | interventions — Acclimatization

STUDY DESIGN:
Intervention Model Description: 80 parents (40 depressed; 40 non-depressed) and their children with EBD will be recruited to complete an assessment to determine objective emotional, cognitive, and behavioural markers. A subset of 20-40 depressed parents who meet inclusion criteria will be recruited for group treatment.
  The aim is to recruit 6-8 parents (and their co-parents) per group for each of 3 consecutive groups (target n = 36). These parents will be invited to participate in 2 individual and 8 weekly group treatment sessions. Following treatment, parents will be invited to a post-group assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Group Treatment (Experimental): Families who meet inclusion criteria will participate in the Parent Group Treatment (ADAPT Program).
  Interventions: Behavioral: Addressing Depression and Positive Parenting Techniques (ADAPT) Program
- No Treatment (No Intervention): Families who do not meet inclusion criteria will not be invited to participate in the ADAPT Program.

INTERVENTIONS:
Behavioral: Addressing Depression and Positive Parenting Techniques (ADAPT) Program — The intervention is a targeted parenting intervention that has modules that help parents build emotion regulation skills, distress tolerance skills and alternative and more helpful ways of thinking about the causes of their child's EBD. The program also includes behavioral parent training skills building modules.
  Arms: Parent Group Treatment

SUMMARY:
Children with emotional and behavioural difficulties (EBD) experience disproportionate social, family and academic impairment and have between two to five times increased likelihood of developing an anxiety disorder, mood disorder or other severe mental illness in adolescence and adulthood. There is a close association between parental depression and the emergence and maintenance of childhood EBD that is likely bidirectional. Parents of children with EBD experience disproportionate stress, increasing their risk for depression; yet chronic and untreated parental depression is associated with the emergence of child EBD in the first place. Therefore, designing targeted and effective assessment and treatment for parents of children with EBD that take into account parents' depression is necessary. Of pressing concern, first-line Behavioral Parent Training (BPT) treatments for parents of children with EBD are not tailored to parent's mental health needs, which may be why upwards of 40 percent of parents and children treated in these programs fail to sufficiently benefit. Existing research highlights emotional and cognitive factors that may differentiate depressed parents from non-depressed parents that may be treatment targets to improve outcomes for depressed parents and children.

The main aim of the proposed project is to evaluate the feasibility and acceptability of a novel targeted treatment for depressed parents of children with EBD, along with adherence to study protocol. The investigators will use the results of the pilot study to make key modifications to study procedures and the treatment itself to increase the success of a future randomized controlled trial (RCT) to test treatment efficacy.

The investigators hypothesize that:

1. Recruitment will be feasible.
2. The intervention will be acceptable, and there will be a high rate of adherence to study protocol.

DETAILED DESCRIPTION:
Study Rationale:

Developmental theories underscore the reciprocal nature of parent-child interactions and the importance of adult teaching and modeling to enable the development of children's emotion regulation, frustration tolerance and behavioural regulation skills. Similarly, these models are bidirectional in that children's skills develop along with, and influence parental cognitions, emotional functioning and the manner in which parent's impose expectations and respond to children's behaviour. Indeed, adult-child transactions can serve to increase or decrease a child and parent's frustration and arousal, fuel response biases in the child and parent, and lead to adaptive or maladaptive parent and child behaviour. Much literature has documented the close association between parental depression and the emergence and maintenance of childhood EBD. From transactional and biopsychosocial perspectives, it has been suggested that depression negatively impacts a parent's ability to regulate their own emotions and cognitions, and subsequently positively attend to their child. As such, parental depression may indirectly contribute to a cycle of behavioural escalation on the part of the child to get their needs met. This is not to suggest that parental depression causes childhood EBD; however, shared genetic and environmental factors may contribute to challenges with parent and child co-regulation of emotion, elevated irritability, unhelpful thinking patterns, and perpetuation of a problematic cycle of interactions. Transactional theory suggests that the "fit" between parental emotional functioning, cognition and behaviour with child emotional and behavioural functioning may be of primary importance, rather than indicating any one ideal parenting approach as is suggested by standard BPT. The transactional model suggests that compatibility between adult and child characteristics and behaviour will produce optimal outcomes. Indeed, the goal of BPT is to help parents develop skills that meet the needs of children with EBD. Current programs may not have sufficient therapeutic components that match the emotional, cognitive and behavioural needs of parents with depression suggesting that alternative and targeted models may be indicated for these parents.

Research Questions:

The aim of the research is to determine the feasibility of novel assessment and treatment for parents with depression that builds parent's functional cognitions, emotion regulation, parenting competencies and skills (Addressing Depression and Positive Parenting Techniques (ADAPT)).

1. To determine the feasibility of recruitment

   1. What is the rate of eligible parents in each of the pilot recruitment sites and overall?
   2. What is parents' level of readiness to engage in parenting treatment?
   3. What is the recruitment rate in each setting and what are reasons for non-participation?
2. To determine feasibility and acceptability of a novel treatment.

   1. What are participant (and clinician) views of the intervention?
   2. What is the rate of completion of the intervention and reasons for discontinuation?
   3. What is the average number of groups attended?
3. Adherence to study protocol

   1. What is the level of clinician adherence to the ADAPT protocol?
   2. What is the follow-up rate for outcome data collection, including measures of parental depression, parenting stress, parenting skills, parent-child interactions and child EBD?

The investigators hypothesize that recruitment will be feasible, that the intervention will be acceptable, and that there will be a high rate of adherence to the study protocol.

Significance of the Study:

Although parents are clearly critically important to the success of BPT, very little research has focused on understanding key parental factors that may be important to assess or on the effectiveness of BPT tailored to parents with depression. Existing research has primarily focused on logistical barriers to treatment such as socioeconomic status or child-factors, such as the severity or type of EBD, that may moderate or mediate BPT outcomes. Important parental factors associated with depression, such as parental cognitions, and parental emotional and behavioural regulation skills, have largely been ignored when designing novel interventions. Systematically understanding differences between parents with and without depression on these key factors and the feasibility of novel treatment will identify avenues for treatment innovation.

Study Design

Clinic-referred parents with depression who have children with EBD will be recruited from the Mood and Anxiety Service (MAAS) Clinic at the Centre for Addiction and Mental Health (CAMH) and the Women's Mental Health Program at Women's College Hospital (WCH). Non-depressed parents of children with EBD will be recruited from the Child, Youth and Emerging Adult Program (CYEAP) at CAMH. The target sample size is 80 parents (40 depressed, 40 non-depressed) and their children with EBD. Participants will be recruited over two years. A multi-modal measurement approach incorporating subjective and objective measures and tasks will be used.

Parent and child psychopathology and treatment outcome will be measured by widely used and validated parent and child-completed interviews, questionnaires and recorded tasks. Measures were chosen based on their sound psychometric properties. Additionally, many of the child-based measures have been used by the PI in ongoing clinical research projects and parent measures used in the MAAS. As such, the feasibility of completing these measures in the clinical setting has been confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Parent is over the age of 18 years and has a child between the ages of 6 and 10;
* Parent shows clinical elevations for Depression on the Patient Health Questionnaire (PHQ);
* The child has clinically elevated Emotional Behavioural Difficulties (T-score of 65, Borderline range, 93rd percentile) on the Strength and Difficulties Questionnaire (Conduct Problem or Total Difficulties subscales);
* The parent's has capacity to tolerate a group context.

Exclusion Criteria:

* Parent shows active suicidal ideation, substance use disorder, or psychosis;
* Parent is not suitable for group treatment based on clinical interview;
* Parent cannot communicate in English;
* Child has a diagnosis of Autism Spectrum Disorder or Intellectual Disability (based on parent report).

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of treatment sessions attended by parents measured using weekly attendance log | 2 years
  Attendance Log - Clinicians leading the group sessions will track session attendance on a weekly basis along with documenting reasons for absenteeism. Treatment/recruitment will be considered feasible if greater than 70 percent of parents attend more than 70 percent of the sessions in each pilot group.
Treatment acceptability/satisfaction measured by weekly evaluation forms filled out by parents | 2 years
  Weekly Evaluation Forms - Participants will be asked to share their opinions about session content and delivery on a weekly basis. The treatment will be considered acceptable if greater than 70 percent of all participants report adequate acceptability of the group treatment.
Clinician adherence to ADAPT protocol measured by fidelity checks | 2 years
  Trained research staff will conduct weekly fidelity checks at the group treatment sessions to track clinician adherence to treatment content. The treatment will be considered acceptable if greater than 70 percent clinician adherence to the model is assessed by review of coded sessions checklists.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan F Andrade, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lundahl B, Risser HJ, Lovejoy MC. A meta-analysis of parent training: moderators and follow-up effects. Clin Psychol Rev. 2006 Jan;26(1):86-104. doi: 10.1016/j.cpr.2005.07.004. Epub 2005 Nov 8. PMID 16280191
- [Background] Luoma I, Tamminen T, Kaukonen P, Laippala P, Puura K, Salmelin R, Almqvist F. Longitudinal study of maternal depressive symptoms and child well-being. J Am Acad Child Adolesc Psychiatry. 2001 Dec;40(12):1367-74. doi: 10.1097/00004583-200112000-00006. PMID 11765281
- [Background] Ludmer JA, Salsbury D, Suarez J, Andrade BF. Accounting for the impact of parent internalizing symptoms on Parent Training benefits: The role of positive parenting. Behav Res Ther. 2017 Oct;97:252-258. doi: 10.1016/j.brat.2017.08.012. Epub 2017 Aug 23. PMID 28863289
- [Background] Aitken M, Waxman JA, MacDonald K, Andrade BF. Effect of Comorbid Psychopathology and Conduct Problem Severity on Response to a Multi-component Intervention for Childhood Disruptive Behavior. Child Psychiatry Hum Dev. 2018 Dec;49(6):853-864. doi: 10.1007/s10578-018-0800-1. PMID 29594940
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Eyberg, S.M., et al. Manual for the dyadic parent-child interaction coding system: Third edition. 2009, University of Florida.
- [Background] Fanti, KA, Panaylotou G, and Fanti S. Associating parental to child psychological symptoms: Investigating a transactional model of development. Journal of Emotional and Behavioral Disorders 21(3): 193-210, 2013.
- [Background] Peris TS, Hinshaw SP. Family dynamics and preadolescent girls with ADHD: the relationship between expressed emotion, ADHD symptomatology, and comorbid disruptive behavior. J Child Psychol Psychiatry. 2003 Nov;44(8):1177-90. doi: 10.1111/1469-7610.00199. PMID 14626458
- [Background] Harvey P, Penzo JA. Parenting a child who has intense emotions: Dialectical behavior therapy skills to help your child regulate emotional outbursts & aggressive behaviors. Oakland, CA: New Harbinger Publications, 2009.
- [Background] Perepletchikova F, Nathanson D, Axelrod SR, Merrill C, Walker A, Grossman M, Rebeta J, Scahill L, Kaufman J, Flye B, Mauer E, Walkup J. Randomized Clinical Trial of Dialectical Behavior Therapy for Preadolescent Children With Disruptive Mood Dysregulation Disorder: Feasibility and Outcomes. J Am Acad Child Adolesc Psychiatry. 2017 Oct;56(10):832-840. doi: 10.1016/j.jaac.2017.07.789. Epub 2017 Aug 10. PMID 28942805